CLINICAL TRIAL: NCT06374004
Title: The Effect of Thoracic Mobilization on Pain Intensity, Muscle Tone, Functional and Muscle Activity Level in Individuals With Subacromial Pain Syndrome
Brief Title: The Effect of Thoracic Mobilization in Individuals With Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mahmut Çalık, MSc, PhD Student, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-FTR-MC-01
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Subacromial Pain Syndrome
Keywords: Rehabilitation; Electromyography; Acromiohumeral Distance; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: One group received exercise therapy and the other group received manual therapy (thoracic mobilization) in addition to exercise therapy
Who Masked: Participant
Masking Description: Participants will be randomly divided into two groups and participants will not know which group participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): The exercise group will perform stretching and strengthening exercises involving the muscle groups around the shoulder and scapula for 12 weeks.
  Interventions: Other: Exercise Group
- Thoracic Mobilization Group (Active Comparator): The exercise group will perform stretching and strengthening exercises involving the muscle groups around the shoulder and scapula for 12 weeks. In addition to the exercises, thoracic mobilization will be applied to the participants in this group 1 day a week for a total of 6 weeks.
  Interventions: Other: Exercise Group; Other: Thoracic Mobilization Group

INTERVENTIONS:
Other: Exercise Group — The exercises will be given as a home program and each exercise will be performed 2 times a day for a total of 12 weeks. Participants will perform the exercises 1 day a week under the supervision of a physiotherapist. The exercise program lasts approximately 30 minutes.
Other: Thoracic Mobilization Group — The exercises will be given as a home program and each exercise will be performed 2 times a day for a total of 12 weeks. Participants will perform the exercises 1 day a week under the supervision of a physiotherapist. The exercise program lasts approximately 30 minutes. Thoracic mobilization will be applied to segments where passive accessory movement is insufficient or painful. 30 repetitions/4 sets will be applied to each determined segment. Thoracic mobilization will be performed with the patient lying prone position.
  Arms: Thoracic Mobilization Group

SUMMARY:
The purpose of this study is to investigate the effect of six-week thoracic mobilization on pain intensity, muscle tone, functional and muscle activation in individuals with subacromial pain syndrome.

DETAILED DESCRIPTION:
Subacromial pain syndrome (SAPS) is the most common shoulder problem and accounts for 44%-65% of all shoulder problems. Repetitive compression of the rotator cuff tendons as they pass through the subacromial space affects shoulder function along with pain.

Studies have shown that scapular kinematics are affected in individuals with subacromial pain syndrome. In addition to increased scapular internal rotation, scapular upward rotation and posterior tilt during elevation are decreased in these individuals. These kinematic changes have been associated with decreased activation of the middle and lower trapezius and serratus anterior muscles and excessive upper trapezius activation. This change in scapular kinematics causes narrowing of the subacromial space and repeated traumatization of the rotator cuff muscles passing through it. In addition, kyphotic posture in the thoracic region (insufficient extension of the thoracic vertebrae) negatively affects scapular kinematics. Kyphotic posture has been shown to be associated with subacromial pain syndrome by causing anterior tilt, downward rotation and protraction in the scapula.

Exercise and mobilization applications are frequently applied in subacromial pain syndrome. Strengthening the muscles around the shoulder and scapula, increasing glenohumeral and scapulothoracic joint mobility, and stretching the posterior capsule are frequently applied to reduce pain and increase function. Studies on increasing thoracic mobilization are limited in number. In these studies, the acute effects of thoracic manipulation applications on pain, normal joint motion and functional activity level were examined in individuals with subacromial pain syndrome. There is only one pilot study that examined the effect of mobilization applied to the thoracic region. The purpose of this study is to investigate the effect of six-week thoracic mobilization on pain intensity, muscle tone, functional and muscle activation in individuals with subacromial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic kyphosis angle > 40°
* Full active shoulder abduction

Exclusion Criteria:

* Bilateral shoulder pain
* Rotator cuff tear
* Shoulder/cervical injury other than SAPS
* Surgery history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Electromyography (EMG) | twelve weeks
  A surface EMG system with 8 channels will use to measure muscle activation levels. A synchronized video record will take at 50 frames per second to identify 3 phases of the exercises ascending phase of the abduction (from 0°-60°, 60°-120°, and 120°-180°). Measurements will make from the affected side. The same examiner will place bipolar Ag-Cl surface electrodes over the Upper Trapezius (UT), Middle Trapezius (MT), Lower Trapezius (LT), Infraspinatus (IS), Middle Deltoid (MD), and Serratus Anterior (SA) muscles of all participants. Investigators will measure maximal voluntary isometric contractions (MVICs) of the UT, MT, LT, IS, MD, and SA muscles in randomized order first.
  The width of the wooden blocks will adjust according to the arm distance of the patients. Shoulder abduction angles of 60° and 120° will mark with tape on the wooden blocks.
Acromiohumeral Distance (AHD) | twelve weeks
  Real-time ultrasonography (US) images of the subacromial space will obtain with a 4 to 13 Megahertz linear transducer. All US images will evaluate by the same researcher with 5 years of experience in US imaging of the shoulder. US images will obtain from the affected side shoulder.
  The AHD will measure linearly (as a millimetres) between the highest point of the humeral head and the lowest point of the acromion using the on-screen calibrations of the US system. Measurements will do at 0°, 60° and 90° abduction of the shoulder.

SECONDARY OUTCOMES:
Muscle Tone | twelve weeks
  The participant's upper trapezius muscle tone will assess. Measurements will make by placing the tip of the muscle tone assessment device vertically at the midpoint of the individuals' upper trapezius muscle. The resulting changes in muscle tone and stiffness will record as results.
Functional Activity Level | twelve weeks
  American Shoulder and Elbow Surgeons (ASES) will use to determine functional activity level. ASES is frequently use in the evaluation of shoulder functions in rotator cuff injuries. Participants can score between 0-100 points in the ASES assessment. A high score on the ASES assessment indicates high activity level and low disability level.The Turkish version of the questionnaire will use in our study.
Pain Intensity | twelve weeks
  A pain intensity will evaluate with the Visual Analog Scale (VAS). Participants will ask to mark the intensity of pain participants feel during rest and night pain and daily life activity on a 0-10 cm straight line. The length between the point will mark by the patient and the starting point on the line will measure with a ruler and the pain intensity will record in cm.

CONTACTS AND LOCATIONS:
Overall Officials: MAHMUT ÇALIK, PhD Student, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)